CLINICAL TRIAL: NCT02084043
Title: In Vitro Comparison of Continuous and Breath-synchronized Vibrating Mesh Nebulizer During Non Invasive Ventilation: Analysis of Inhaled and Lost Doses.
Brief Title: In Vitro Assessment of a Breath-synchronized Vibrating Mesh Nebulizer During Non Invasive Ventilation
Acronym: Synchro-Neb
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital St Luc, Brussels (Other)
Collaborators: Université Catholique de Louvain (Other); University of Applied Sciences of Western Switzerland (Other); School of Gestion and Engineering Vaud, Switzerland (Unknown)
Responsible Party: Principal Investigator, Jean-Bernard Michotte, MSc, PhD Student, University of Applied Sciences of Western Switzerland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Synchro-Neb
Record Dates: First submitted 2014-03-08; First posted 2014-03-11 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Respiratory Diseases; Lung Diseases; Cystic Fibrosis; COPD; Asthma
Keywords: aerosol delivery; vibrating mesh nebulizer; breath-actuated nebulizer; non invasive ventilation; bilevel ventilator; single limb circuit ventilator; Amikacin
MeSH Terms: conditions — Respiratory Tract Diseases; Lung Diseases; Cystic Fibrosis; Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Breath-actuated vibrating mesh nebulizer (Experimental): 500 mg/4 mL of Amikacin solution delivered with an experimental breath-actuated vibrating mesh nebulizer associated with a single limb circuit ventilator.
  Interventions: Drug: Nebulization of Amikacin during NIV (RR: 15 cycles/minute); Drug: Nebulization of Amikacin during NIV (RR: 25 cycles/minute)
- Conventional vibrating mesh nebulizer (Experimental): 500 mg/4 mL of Amikacin solution delivered with a conventional vibrating mesh nebulizer (in continuous mode) associated with a single limb circuit ventilator.
  Interventions: Drug: Nebulization of Amikacin during NIV (RR: 15 cycles/minute); Drug: Nebulization of Amikacin during NIV (RR: 25 cycles/minute)

INTERVENTIONS:
Drug: Nebulization of Amikacin during NIV (RR: 15 cycles/minute) — 500 mg/4 mL Amikacin nebulized using vibrating mesh nebulizer associated with a single limb bilevel ventilator. The nebulizations are considered as finished when there is no visible evidence of nebulization for a period of 30 seconds. The NIV is set with an IPAP of 15 cmH2O and EPAP of 5 cmH2O. The lung model is simulated with a respiratory rate of 15 cycles/minute
  Other Names: Amikacine sulfate
Drug: Nebulization of Amikacin during NIV (RR: 25 cycles/minute) — 500 mg/4 mL Amikacin nebulized using vibrating mesh nebulizer associated with a single limb bilevel ventilator. The nebulizations are considered as finished when there is no visible evidence of nebulization for a period of 30 seconds. The NIV is set with an IPAP of 15 cmH2O and EPAP of 5 cmH2O. The lung model is simulated with a respiratory rate of 25 cycles/minute
  Other Names: Amikacine sulfate

SUMMARY:
Using an adult lung bench model of non invasive ventilation, the aim of the study is to compare an experimental system of breath-synchronized vibrating mesh nebulizer to a conventional vibrating mesh nebulizer during non invasive ventilation in terms of inhaled and lost doses.

ELIGIBILITY:
Inclusion Criteria:

* Not applicable (in vitro study)

Exclusion Criteria:

* hypersensitivity (allergic) reactions to aminoglycosides

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Inhaled dose | after 24 hours
  The inhaled dose assessed by residual gravimetric method

SECONDARY OUTCOMES:
Expiratory wasted dose | after 24 hours
  The dose expelled in the ambient air through the exhalation port assessed by residual gravimetric method

OTHER OUTCOMES:
Estimated lost dose | after 24 hours
  The dose lost into the circuit (nebulizer included) assessed by residual gravimetric method

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Bernard Michotte, PhD student, Principal Investigator — University of Health Sciences (HESAV); Jonathan Dugernier, PhD student, Principal Investigator — Cliniques universitaires Saint-Luc, service des soins intensifs; Enrico Staderini, PhD, Principal Investigator — School of Gestion and Engineering Vaud (HEIG-VD); Rares Rusu, MSc, Study Chair — School of Gestion and Engineering Vaud (HEIG-VD); Jean Roeseler, PhD, Study Chair — Cliniques universitaires Saint-Luc, service des soins intensifs; Giuseppe Liistro, MD PhD, Study Chair — Cliniques universitaires Saint-Luc, service de pneumologie; Gregory Reychler, PhD, Study Director — Cliniques universitaires Saint-Luc, service de pneumologie
Locations (1):
- University Hospital St Luc, Brussels, Belgium